CLINICAL TRIAL: NCT01369914
Title: The Natural History of Ocular Graft-Versus Host Disease
Brief Title: The Natural History of Graft-Versus-Host Disease in the Eyes
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110173; 11-EI-0173
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2016-02-05

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft-Versus-Host Disease; Natural History Study; Hematopoietic Stem Cell Transplant; GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Background:

* Stem cell transplantation (SCT) is used to treat some kinds of cancer, blood cell disorders, and immune disorders. Stem cells from a donor s blood are used to replace the recipient s stem cells in the bone marrow. The recipient s bone marrow can then produce new blood cells. Some of these new cells involved in the immune system are like the donor s cells. Sometimes immune cells from the SCT attack the recipient s normal tissues, including the eyes. This type of immune attack is called graft-versus-host disease, or GVHD.
* The symptoms of ocular GVHD include eye pain, irritation, dryness, and inflammation. When it is severe and if it does not respond well to treatment, ocular GVHD may also cause vision loss.

Objective:

- To learn more about graft-versus-host disease (GVHD) of the eyes in people who have had stem cell transplantation.

Eligibility:

* Participants must be at least 18 years of age.
* They must be taking part in a study at the National Cancer Institute (NCI) or the National Heart, Lung and Blood Institute (NHLBI).
* They must have a SCT scheduled within the next 30 days.

Design:

* The study lasts for 1 year and includes six visits to the National Eye Institute. (There is an optional visit about 1 month before your SCT.) When possible, visits for this study will be scheduled so that they can be done on the same day as your visits for the NCI or NHLBI protocol that you are taking part in.
* At each visit, participants will have a medical exam and an eye history will be taken. They will have an eye exam and a test to measure the ability to make tears. Those in the study will also have tear fluid collected for analysis in a lab. Tear fluid collection is a painless process. Blood will be drawn during certain visits if it has not already been collected by the transplant team.

DETAILED DESCRIPTION:
OBJECTIVE:

The study objectives are to study the development of ocular graft-versus-host disease (GVHD) in participants treated with stem cell transplantation (SCT) at the NIH, including exam findings prior to SCT, changes in ocular signs and symptoms following SCT and response to standard therapy in participants identified with dry eye and ocular GVHD; to develop clinical outcome measures for early onset and more advanced ocular GVHD and provide estimates of progression rates for these outcomes; to analyze tear fluid, impression cytology (IC) and serum samples from participants undergoing SCT, to identify biomarkers or other findings which may predict the onset of ocular GVHD or correlate with disease progression or response to therapy and to establish a cohort of participants with ocular GVHD in anticipation of future clinical trials.

STUDY POPULATION:

Up to 50 adult participants undergoing SCT at the NIH, and up to 50 healthy adult participants will be enrolled.

DESIGN:

This prospective, natural history study will follow participants through 12 months post-SC, with the option to extend follow-up for up to five years.

OUTCOME MEASURES:

The primary objective outcome variable is ocular surface staining using fluorescein and lissamine green dyes, as measured by the Oxford criteria, with the scale ranging from 0 to 15 in each eye. The primary subjective outcome measure is the Ocular Surface Disease Index (OSDI), ranging from 0 to 100. Secondary outcome variables include best-corrected visual acuity (BCVA), tear film osmolarity, Schirmer s tear testing with anesthesia, meibomian gland function and tear break-up time. In addition, tear fluid biomarkers and/or IC will be studied as secondary outcome variables to determine whether changes in biomarker levels (tear fluid) or cell densities and morphologies (IC) correlate with the development or progression of ocular GVHD.

ELIGIBILITY:
* INCLUSION CRITERIA:

SCT Participants

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol s informed consent document.
3. Participant is scheduled for a SCT under another NIH protocol within the next 30 days.
4. Participant is willing and able to comply with the study procedures and follow-up visits.

Healthy Participants

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol s informed consent document.
3. Participant has no more than minimal current dry eye disease, defined as no more than minimal dry eye symptoms, Schirmer s with anesthesia (Bullet) 6, tear break-up time (TBUT) (Bullet) 6, and corneal staining (Oxford) < 3 in both eyes.

EXCLUSION CRITERIA:

SCT Participants

1. Participant has a history of ocular problems which could interfere with the natural history of their response to treatment with SCT. Examples include significant dry eye disease, use of cyclosporine eye drops in the past 30 days and conjunctival scarring for any reason.
2. Participant has known allergies to dilating or anesthetic eye drops.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-05-20; Study Completion 2016-02-05

PRIMARY OUTCOMES:
The primary objective variable is ocular surface staining using fluorescein and lissamine green dyes. The primary subjective outcome measure is the OSDI | Ongoing

SECONDARY OUTCOMES:
In addition, tear fluid biomarkers and conjunctival IC will be studied as a secondary outcome variable to determine whether changes in biomarker levels or cell densities and morphologies correlate with the development or progression of ocular GV... | Ongoing
Secondary outcome variables include changes in BCVA (ETDRS); tear film osmolarity; Schirmer's testing with anesthesia; meibomain gland function; tear break-up time. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Rachel J Bishop, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Jabs DA, Wingard J, Green WR, Farmer ER, Vogelsang G, Saral R. The eye in bone marrow transplantation. III. Conjunctival graft-vs-host disease. Arch Ophthalmol. 1989 Sep;107(9):1343-8. doi: 10.1001/archopht.1989.01070020413046. PMID 2675805
- [Background] Kim SK. Update on ocular graft versus host disease. Curr Opin Ophthalmol. 2006 Aug;17(4):344-8. doi: 10.1097/01.icu.0000233952.09595.d8. PMID 16900025